CLINICAL TRIAL: NCT02949921
Title: Radiesse® Post Approval Safety Study - Radiological Evaluation of Implantation in the Hands
Brief Title: Radiological Evaluation of Radiesse Implantation in the Hands
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P151010, M900311003
Record Dates: First submitted 2016-09-13; First posted 2016-10-31 (Estimated); Results first posted 2019-03-14 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Volume Loss in the Dorsum of the Hand

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- "Grade 4 Hands" group (Experimental): "Grade 4 Hands" group will be subjects with hand grading of grade 4 (very severe loss of fatty tissue, marked visibility of veins and tendons in the dorsal hand). "Grade 4 Hands" group subjects will receive Radiesse injectable implant and 2% lidocaine HCL up to 3 cc (2 syringes) per hand per treatment. Subjects in "Grade 4 Hands" group can have up to three retreatments over an 18 month period.
  Interventions: Device: Radiesse injectable implant and 2% lidocaine HCL
- "Grade 2 or 3 Hands" group (Experimental): "Grade 2 or 3 Hands" group will be subjects with hand grading of grade 2 or grade 3 (moderate to severe loss of fatty tissue, mild to moderate visibility of veins and tendons in the dorsal hand). "Grade 2 or 3 Hands" group subjects will receive Radiesse injectable implant and 2% lidocaine HCL up to 3 cc (2 syringes) per hand per treatment. Subjects in "Grade 2 or 3 Hands" group can have up to three retreatments over an 18 month period.
  Interventions: Device: Radiesse injectable implant and 2% lidocaine HCL

INTERVENTIONS:
Device: Radiesse injectable implant and 2% lidocaine HCL — Radiesse injectable implant injected in small boluses (0.2-0.5cc/bolus). No more than 0.5cc per bolus. No more than 3 cc (2 syringes) will be injected per hand.

SUMMARY:
The objective of this study is to provide a preliminary assessment of the radiographic appearance of Radiesse material that has been injected into the dorsum of the hands.

DETAILED DESCRIPTION:
Radiesse dermal filler is radiopaque and shows no overt radiographic safety concerns in a study of 58 patients after facial implantation, with Radiesse not always visible on plain X-rays.

This Post Approval Safety study will evaluate if there are concerns after Radiesse implantation in the dorsum of hands, specifically if implantation interferes with radiological assessment by obscuring the bones of the hand.

Hands will be scored according to the 5 point Merz Hand Grading Scale (MHGS), which ranges from 0 (No loss of fatty tissue) to 4 (Very severe loss of fatty tissue; marked visibility of veins and tendons).

ELIGIBILITY:
Inclusion Criteria:

1. Has hands rating 2, 3, or 4 on the validated Merz Hand Grading Scale (MHGS) as determined by a live, masked evaluator.
2. Is at least 22 years of age.
3. Understands and accepts the obligation not to receive any other procedures in the dorsum of the hands through the end of the study.

Exclusion Criteria:

1. Was a participant in the Radiesse hands pre-market clinical study.
2. Has been treated with fat injections or Radiesse in the hands, has hand deformities, or has received surgery in the dorsum of the hands.
3. Has any medical condition with the potential to interfere with the study or increase the risk of adverse events (AEs).

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2018-01-02 (Actual); Study Completion 2018-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kreymerman, MD,FACS, Study Director — Study Director
Locations (1):
- Merz Investigative Site #0010358, Vista, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moradi A, Ethakovic R, Odena G. Aesthetic Implantation of Calcium Hydroxylapatite Does Not Interfere With Radiological Assessment of Bones in the Dorsum of the Hands. Aesthet Surg J. 2023 May 15;43(6):696-703. doi: 10.1093/asj/sjac344. PMID 36573029

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 1 investigative site in the United States.
Pre-assignment Details: A total of 20 participants were enrolled, treated, and completed the study.
Groups:
- Group A: MHGS Grade 4 Hands Group: Participants with Merz hand grading scale (MHGS) Grade 4, which indicates very severe loss of fatty tissue, marked visibility of veins and tendons in the dorsal hand, received Radiesse injectable implant and 2 percent (%) lidocaine hydrochloric acid (HCL) up to 3 cubic centimeter (cc) (2 syringes) per hand per treatment on Day 7 (Week 1). All participants were treated in the dorsum of the hands. Based on the investigator and participant's decision, participants received up to three retreatments at Months 6, 12, and 18.
- Group B: MHGS Grade 2 or 3 Hands Group: Participants with MHGS Grade 2 or 3, which indicates moderate to severe loss of fatty tissue, mild to moderately visibility of veins and tendons in the dorsal hand, received Radiesse injectable implant and 2% lidocaine HCL up to 3 cc (2 syringes) per hand per treatment on Day 7 (Week 1). All participants were treated in the dorsum of the hands. Based on the investigator and participant's decision, participants received up to three retreatments at Months 6, 12, and 18.
Period: Overall Study
Arm/Group | Group A: MHGS Grade 4 Hands Group | Group B: MHGS Grade 2 or 3 Hands Group
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who were enrolled in the study.
Groups:
- Group A: MHGS Grade 4 Hands Group: Participants with MHGS Grade 4, which indicates very severe loss of fatty tissue, marked visibility of veins and tendons in the dorsal hand, received Radiesse injectable implant and 2% lidocaine HCL up to 3 cc (2 syringes) per hand per treatment on Day 7 (Week 1). All participants were treated in the dorsum of the hands. Based on the investigator and participant's decision, participants received up to three retreatments at Months 6, 12, and 18.
- Total: Total of all reporting groups
Arm/Group | Group A: MHGS Grade 4 Hands Group | Group B: MHGS Grade 2 or 3 Hands Group | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (7.40) | 53.3 (9.83) | 57.5 (9.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 9 | 9 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 10 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — Skin type I = white; very fair, red or blonde hair blue eyes; freckles; always burns, never tans, skin type II = white, fair, red or blond hair; blue, hazel or green eyes; usually burns, tans with difficulty, skin type III = cream white; fair with any eye or hair color (common); sometimes mild burn, gradually tans, skin type IV = brown; typical Mediterranean Caucasian skin; rarely burns, tans with ease, skin type V = dark brown; mid-eastern skin types; very rarely burns, tans easily, and skin type VI = black; never burns, tans very easily.
  Participants
    Skin Type I | 0 | 0 | 0
    Skin Type II | 6 | 4 | 10
    Skin Type III | 3 | 6 | 9
    Skin Type IV | 1 | 0 | 1
    Skin Type V | 0 | 0 | 0
    Skin Type VI | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With X-ray of Either Hand With Bone Obscuration at Month 1
Description: Obscuration was defined as any post-treatment hand x-ray that at least 1 of the 2 blinded radiologist interpreted as Radiesse obscuring bones.
Time Frame: Month 1
Population: All participants who were enrolled in the study.
Measure: Number; unit: participants
Arm/Group | Group A: MHGS Grade 4 Hands Group | Group B: MHGS Grade 2 or 3 Hands Group
Number analyzed (Participants) | 10 | 10
participants | 0 | 0

2. Primary Outcome: Number of Participants With X-ray of Either Hand With Bone Obscuration at Month 6
Description: as for outcome 1
Time Frame: Month 6
Population: All participants who were enrolled in the study.
Measure: Number; unit: participants
Arm/Group | Group A: MHGS Grade 4 Hands Group | Group B: MHGS Grade 2 or 3 Hands Group
Number analyzed (Participants) | 10 | 10
participants | 0 | 0

3. Primary Outcome: Number of Participants With X-ray of Either Hand With Bone Obscuration at Month 12
Description: as for outcome 1
Time Frame: Month 12
Population: Data was not calculated since no participant had bone obscuration at Month 6, and therefore no x-ray was taken at Month 12.
Arm/Group | Group A: MHGS Grade 4 Hands Group | Group B: MHGS Grade 2 or 3 Hands Group
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Number of Participants With X-ray of Either Hand With Bone Obscuration at Month 24
Description: as for outcome 1
Time Frame: Month 24
Population: Participants who received 4 treatments in total (initial and 3 retreatments).
Measure: Number; unit: participants
Arm/Group | Group A: MHGS Grade 4 Hands Group | Group B: MHGS Grade 2 or 3 Hands Group
Number analyzed (Participants) | 4 | 2
participants | 0 | 0

5. Secondary Outcome: Percentage of Participants Reporting One or More Device or Injection-related Severe Adverse Events (AEs) at Months 1 and 6
Time Frame: Months 1 and 6
Population: All participants who were enrolled in the study.
Measure: Number; unit: percentage of participants
Arm/Group | Group A: MHGS Grade 4 Hands Group | Group B: MHGS Grade 2 or 3 Hands Group
Number analyzed (Participants) | 10 | 10
percentage of participants
  Month 1 | 0 | 10.0
  Month 6 | 0 | 10.0

6. Secondary Outcome: Michigan Hand Outcomes Questionnaire (MHQ) Scores
Description: The MHQ is a hand-specific outcomes instrument that measures outcomes of participants with conditions of, or injury to, the hand or wrist. The MHQ contains six domains: overall hand function, activities of daily living, work performance, pain, aesthetics and satisfaction. For this study, MHQ overall hand function and MHQ pain domains were evaluated. Scores for both scales range from 0-100. Higher MHQ hand function scores denote better hand performance whereas higher MHQ pain scores denote more pain. MHQ minimal clinically important differences were defined as score changes greater than an 11-point increase for the pain domain and greater than a 13-point decrease for the function domain.
Time Frame: Baseline, Months 1, 6, 7, 12, 13, 18, 19 and 24
Population: All participants who were enrolled in the study. Participants who were evaluable for this measure at given time period were included in the assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group A: MHGS Grade 4 Hands Group | Group B: MHGS Grade 2 or 3 Hands Group
Number analyzed (Participants) | 10 | 10
units on a scale
  Baseline: Left Hand (Function) | 96.5 (6.69) | 94.0 (12.87)
  Baseline: Left Hand (Pain) | 2.0 (4.83) | 4.0 (8.10)
  Baseline: Right Hand (Function) | 99.0 (3.16) | 96.5 (6.69)
  Baseline: Right Hand (Pain) | 1.0 (2.11) | 3.5 (8.18)
  Month 1: Left Hand (Function) | 99.5 (1.58) | 98.5 (4.74)
  Month 1: Left Hand (Pain) | 4.5 (6.43) | 4.5 (11.17)
  Month 1: Right Hand (Function) | 99.5 (1.58) | 97.5 (5.40)
  Month 1: Right Hand (Pain) | 2.0 (3.50) | 4.5 (9.56)
  Month 6: Left Hand (Function) | 98.5 (4.74) | 100.0 (0.00)
  Month 6: Left Hand (Pain) | 0.5 (1.58) | 0.0 (0.00)
  Month 6: Right Hand (Function) | 100.0 (0.00) | 100.0 (0.00)
  Month 6: Right Hand (Pain) | 0.0 (0.00) | 0.0 (0.00)
  Month 7: Left Hand (Function): number analyzed (Participants) | 7 | 4
  Month 7: Left Hand (Function) | 99.3 (1.89) | 100.0 (0.00)
  Month 7: Left Hand (Pain): number analyzed (Participants) | 7 | 4
  Month 7: Left Hand (Pain) | 0.0 (0.00) | 0.0 (0.00)
  Month 7: Right Hand (Function): number analyzed (Participants) | 7 | 4
  Month 7: Right Hand (Function) | 100.0 (0.00) | 100.0 (0.00)
  Month 7: Right Hand (Pain): number analyzed (Participants) | 7 | 4
  Month 7: Right Hand (Pain) | 0.0 (0.00) | 0.0 (0.00)
  Month 12: Left Hand (Function) | 99.0 (3.16) | 98.0 (6.32)
  Month 12: Left Hand (Pain) | 0.5 (1.58) | 1.5 (4.74)
  Month 12: Right Hand (Function) | 100.0 (0.00) | 98.0 (6.32)
  Month 12: Right Hand (Pain) | 0.0 (0.00) | 4.5 (14.23)
  Month 13: Left Hand (Function): number analyzed (Participants) | 8 | 8
  Month 13: Left Hand (Function) | 99.4 (1.77) | 100.0 (0.00)
  Month 13: Left Hand (Pain): number analyzed (Participants) | 8 | 8
  Month 13: Left Hand (Pain) | 0.6 (1.77) | 0.0 (0.00)
  Month 13: Right Hand (Function): number analyzed (Participants) | 8 | 8
  Month 13: Right Hand (Function) | 100.0 (0.00) | 100.0 (0.00)
  Month 13: Right Hand (Pain): number analyzed (Participants) | 8 | 8
  Month 13: Right Hand (Pain) | 0.0 (0.00) | 0.0 (0.00)
  Month 18: Left Hand (Function) | 99.5 (1.58) | 100.0 (0.00)
  Month 18: Left Hand (Pain) | 0.5 (1.58) | 0.0 (0.00)
  Month 18: Right Hand (Function) | 100.0 (0.00) | 100.0 (0.00)
  Month 18: Right Hand (Pain) | 0.0 (0.00) | 0.0 (0.00)
  Month 19: Left Hand (Function): number analyzed (Participants) | 7 | 4
  Month 19: Left Hand (Function) | 99.3 (1.89) | 100.0 (0.00)
  Month 19: Left Hand (Pain): number analyzed (Participants) | 7 | 4
  Month 19: Left Hand (Pain) | 0.0 (0.00) | 0.0 (0.00)
  Month 19: Right Hand (Function): number analyzed (Participants) | 7 | 4
  Month 19: Right Hand (Function) | 100.0 (0.00) | 100.0 (0.00)
  Month 19: Right Hand (Pain): number analyzed (Participants) | 7 | 4
  Month 19: Right Hand (Pain) | 0.0 (0.00) | 0.0 (0.00)
  Month 24: Left Hand (Function) | 99.5 (1.58) | 100.0 (0.00)
  Month 24: Left Hand (Pain) | 0.0 (0.00) | 0.0 (0.00)
  Month 24: Right Hand (Function) | 100.0 (0.00) | 100.0 (0.00)
  Month 24: Right Hand (Pain) | 1.0 (3.16) | 0.0 (0.00)

7. Secondary Outcome: Number of Participants With Greater Than or Equal to (>=) 1 Point Improvement on the MHGS in Both Hands After Initial Treatment at Months 1 and 6
Description: The MHGS was used to measure clinical efficacy of the Radiesse hand treatments by a masked evaluator performing live, dorsal hand assessments. The MHGS was an ordinal scale; therefore, ratings were made based on a "snap-shot" at a specific study time point. A measure of successful or improved treatment effect was demonstrated by a decrease in MHGS score. MHGS had 5 categories, where: 0 (no loss of fatty tissue); 1 (mild loss of fatty tissue; slight visibility of veins); 2 (moderate loss of fatty tissue; mild visibility of veins and tendons); 3 (severe loss of fatty tissue; moderate visibility of veins and tendons); 4(very severe loss of fatty tissue; marked visibility of veins and tendons).
Time Frame: Months 1 and 6
Population: All participants who were enrolled in the study.
Measure: Number; unit: participants
Arm/Group | Group A: MHGS Grade 4 Hands Group | Group B: MHGS Grade 2 or 3 Hands Group
Number analyzed (Participants) | 10 | 10
participants
  Month 1 | 10 | 10
  Month 6 | 8 | 9

8. Secondary Outcome: Number of Participants With >=1 Point Improvement on the MHGS in Both Hands Following Retreatment at Months 7 and 12
Description: as for outcome 7
Time Frame: Months 7 and 12
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Group A: MHGS Grade 4 Hands Group | Group B: MHGS Grade 2 or 3 Hands Group
Number analyzed (Participants) | 7 | 4
participants
  Month 7 | 7 | 4
  Month 12 | 5 | 3

9. Secondary Outcome: Percentage of Participants With Global Aesthetic Improvement Scale (GAIS) Scores After Initial Treatment at Months 1 and 6
Description: The GAIS is a 7-point scale. The 7-point scale are as follows: +3 (very much improved); +2 (much improved); +1 (improved); 0 (no change); -1 (worse); -2 (much worse); -3 (very much worse).
Time Frame: Months 1 and 6
Population: All participants who were enrolled in the study.
Measure: Number; unit: percentage of participants
Arm/Group | Group A: MHGS Grade 4 Hands Group | Group B: MHGS Grade 2 or 3 Hands Group
Number analyzed (Participants) | 10 | 10
percentage of participants
  Month 1: Left hand (very much improved) | 60.0 | 60.0
  Month 1: Right hand (very much improved) | 60.0 | 60.0
  Month 1: Left hand (much improved) | 10.0 | 40.0
  Month 1: Right hand (much improved) | 10.0 | 40.0
  Month 1: Left hand (improved) | 30.0 | 0.0
  Month 1: Right hand (improved) | 30.0 | 0.0
  Month 1: Left hand (no change) | 0.0 | 0.0
  Month 1: Right hand (no change) | 0.0 | 0.0
  Month 1: Left hand (worse) | 0.0 | 0.0
  Month 1: Right hand (worse) | 0.0 | 0.0
  Month 1: Left hand (much worse) | 0.0 | 0.0
  Month 1: Right hand (much worse) | 0.0 | 0.0
  Month 1: Left hand (very much worse) | 0.0 | 0.0
  Month 1: Right hand (very much worse) | 0.0 | 0.0
  Month 6: Left hand (very much improved) | 20.0 | 30.0
  Month 6: Right hand (very much improved) | 20.0 | 30.0
  Month 6: Left hand (much improved) | 20.0 | 20.0
  Month 6: Right hand (much improved) | 20.0 | 20.0
  Month 6: Left hand (improved) | 50.0 | 40.0
  Month 6: Right hand (improved) | 50.0 | 40.0
  Month 6: Left hand (no change) | 10.0 | 10.0
  Month 6: Right hand (no change) | 10.0 | 10.0
  Month 6: Left hand (worse) | 0.0 | 0.0
  Month 6: Right hand (worse) | 0.0 | 0.0
  Month 6: Left hand (much worse) | 0.0 | 0.0
  Month 6: Right hand (much worse) | 0.0 | 0.0
  Month 6: Left hand (very much worse) | 0.0 | 0.0
  Month 6: Right hand (very much worse) | 0.0 | 0.0

10. Secondary Outcome: Percentage of Participants With GAIS Scores Following Retreatment at Months 7 and 12
Description: as for outcome 9
Time Frame: Months 7 and 12
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Group A: MHGS Grade 4 Hands Group | Group B: MHGS Grade 2 or 3 Hands Group
Number analyzed (Participants) | 7 | 4
percentage of participants
  Month 7: Left hand (very much improved) | 57.1 | 75.0
  Month 7: Right hand (very much improved) | 57.1 | 75.0
  Month 7: Left hand (much improved) | 28.6 | 0.0
  Month 7: Right hand (much improved) | 28.6 | 0.0
  Month 7: Left hand (improved) | 14.3 | 25.0
  Month 7: Right hand (improved) | 14.3 | 25.0
  Month 7: Left hand (no change) | 0.0 | 0.0
  Month 7: Right hand (no change) | 0.0 | 0.0
  Month 7: Left hand (worse) | 0.0 | 0.0
  Month 7: Right hand (worse) | 0.0 | 0.0
  Month 7: Left hand (much worse) | 0.0 | 0.0
  Month 7: Right hand (much worse) | 0.0 | 0.0
  Month 7: Left hand (very much worse) | 0.0 | 0.0
  Month 7: Right hand (very much worse) | 0.0 | 0.0
  Month 12: Left hand (very much improved) | 28.6 | 25.0
  Month 12: Right hand (very much improved) | 28.6 | 25.0
  Month 12: Left hand (much improved) | 14.3 | 50.0
  Month 12: Right hand (much improved) | 14.3 | 50.0
  Month 12: Left hand (improved) | 42.9 | 0.0
  Month 12: Right hand (improved) | 42.9 | 0.0
  Month 12: Left hand (no change) | 14.3 | 25.0
  Month 12: Right hand (no change) | 14.3 | 25.0
  Month 12: Left hand (worse) | 0.0 | 0.0
  Month 12: Right hand (worse) | 0.0 | 0.0
  Month 12: Left hand (much worse) | 0.0 | 0.0
  Month 12: Right hand (much worse) | 0.0 | 0.0
  Month 12: Left hand (very much worse) | 0.0 | 0.0
  Month 12: Right hand (very much worse) | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: Baseline up to Month 24
Description: The investigator asked the participant for adverse events (AEs) systematically at each visit.
Arm/Group | Group A: MHGS Grade 4 Hands Group | Group B: MHGS Grade 2 or 3 Hands Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 6/10 | 8/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A: MHGS Grade 4 Hands Group (N=10) | Group B: MHGS Grade 2 or 3 Hands Group (N=10)
Nodule (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Swelling (General disorders) | 1 | 3
Herpes zoster (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Animal scratch (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Dental implantation (Surgical and medical procedures) | 1 | 0
Oral surgery (Surgical and medical procedures) | 1 | 0
Rotator cuff repair (Surgical and medical procedures) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of study information usually requires agreement with the sponsor. In case of justified doubts by the sponsor, the INVESTIGATOR will consider these doubts in the publication as long as the scientific neutrality is not affected.

DOCUMENTS (2):
  • Study Protocol (2016-12-13): https://cdn.clinicaltrials.gov/large-docs/21/NCT02949921/Prot_001.pdf
  • Statistical Analysis Plan (2017-04-14): https://cdn.clinicaltrials.gov/large-docs/21/NCT02949921/SAP_000.pdf